CLINICAL TRIAL: NCT04553250
Title: Randomized Controlled Clinical Trial on Lateral Invagination of the Colorectal Anastomosis by Double Stapling
Brief Title: Lateral Invagination of the Colorectal Anastomosis by Double Stapling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Antonio M Lacy, Professor and Head of Gastrointestinal Surgery Department, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2020/1057
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Anastomotic Leak; Sigmoid Diseases
Keywords: anastomotic leak; doubled-stapled anastomosis
MeSH Terms: conditions — Anastomotic Leak; Sigmoid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional technique (Active Comparator): In this group, double-staple colorectal anastomosis will be performed following the technique described by Lee et al: Prior to firing the endostapler, a suture will be placed on the rectal stump that includes both "dog ears". After the punch comes out of the endostapler, the point will be tied, which will invaginate the two corners of the staple line on the same punch. Subsequently, the endostapler will be closed and fired, including the "dog ears" in the anastomotic rims
  Interventions: Procedure: Doubled-stapled colorectal anastomosis
- Lateral invagination technique (Active Comparator): In this group, the circular endostapler will be fired in a conventional way, that is, without having invaginated the two corners of the staple line.
  Interventions: Procedure: Doubled-stapled colorectal anastomosis

INTERVENTIONS:
Procedure: Doubled-stapled colorectal anastomosis — Anastomosis performed between the colon an the rectal stump, using a double-stapled technique.

SUMMARY:
Anastomotic dehiscence is the most feared complication in colorectal surgery, occurring in 6.3% -13.7% in patients with pelvic anastomoses [1-4]. This complication significantly increases morbidity, mortality, costs, and generates a greater impact on quality of life. In addition, several studies point to an increased risk of locoregional recurrence [5, 6].

There are different risk factors for anastomotic dehiscence: some preoperative, such as malnutrition or obesity [9]; other intraoperative ones, such as hypoperfusion of the anastomotic tissue or the anastomotic technique; and others postoperative, such as some types of medication [7]. In colorectal anastomoses, there is some concern about the safety of the double stapling technique, since the extremes of the linear suture line (called "dog ears") and the number of staple lines have a direct relationship with the risk of dehiscence [8-11].

With the aim of reducing suture dehiscence rates, different intraoperative techniques have been developed, such as reinforcing the anastomosis with stitches, the use of indocyanine green [12, 13] or the application of anastomotic sealants [14], without finding a definitive solution. Recently, benefits have been published of using the double-staple colorectal anastomosis lateral invagination technique, with the aim of avoiding "dog ears" [15-17]. Several case series and retrospective comparative studies have shown a significant decrease in anastomotic dehiscence using this technique, with all the clinical and economic benefits that this entails [15-17]. In this sense, the present study aims to evaluate the effectiveness and safety of the lateral invagination technique of double-staple colorectal anastomosis in a randomized and controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Indication of resection of the left colon, sigmoid or upper rectum
* Minimally invasive approach
* Open surgery approach
* Double staple colorectal anastomosis
* Signed informed consent for inclusion in the study

Exclusion Criteria:

* Patients <18 years
* Pregnancy
* ASA> III
* Absolute contraindication for anesthesia
* Patients who receive more than 1 gastrointestinal anastomosis during the same procedure
* Planned multi-organ resection during the same procedure
* Urgent / emergent surgery
* Reinforced anastomosis after positive intraoperative leak test
* Patients with simultaneous application of debulking and HIPEC
* Crohn's disease or active ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 786 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomotic dehiscence diagnosed in the first 30 postoperative days | 30 days
  anastomotic dehiscence diagnosis

SECONDARY OUTCOMES:
Duration of surgery | 1 day
Rate of perioperative morbidity using the Clavien-Dindo classification. | 30 and 90 days PO or in-hospital stay
Rate of perioperative mortality | 30 and 90 days PO or in-hospital stay
Duration of hospital stay | days
Rate of hospital readmissions | 30 days
Rate of surgical reinterventions | 30 days
Rate Stoma closure | 1 year
Rate of Stoma-free survival | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang CY, Halabi WJ, Chaudhry OO, Nguyen V, Pigazzi A, Carmichael JC, Mills S, Stamos MJ. Risk factors for anastomotic leakage after anterior resection for rectal cancer. JAMA Surg. 2013 Jan;148(1):65-71. doi: 10.1001/2013.jamasurg.2. PMID 22986932
- [Background] den Dulk M, Marijnen CA, Collette L, Putter H, Pahlman L, Folkesson J, Bosset JF, Rodel C, Bujko K, van de Velde CJ. Multicentre analysis of oncological and survival outcomes following anastomotic leakage after rectal cancer surgery. Br J Surg. 2009 Sep;96(9):1066-75. doi: 10.1002/bjs.6694. PMID 19672927
- [Background] Peeters KC, Tollenaar RA, Marijnen CA, Klein Kranenbarg E, Steup WH, Wiggers T, Rutten HJ, van de Velde CJ; Dutch Colorectal Cancer Group. Risk factors for anastomotic failure after total mesorectal excision of rectal cancer. Br J Surg. 2005 Feb;92(2):211-6. doi: 10.1002/bjs.4806. PMID 15584062
- [Background] Paun BC, Cassie S, MacLean AR, Dixon E, Buie WD. Postoperative complications following surgery for rectal cancer. Ann Surg. 2010 May;251(5):807-18. doi: 10.1097/SLA.0b013e3181dae4ed. PMID 20395841
- [Background] Senagore A, Lane FR, Lee E, Wexner S, Dujovny N, Sklow B, Rider P, Bonello J; Bioabsorbable Staple Line Reinforcement Study Group. Bioabsorbable staple line reinforcement in restorative proctectomy and anterior resection: a randomized study. Dis Colon Rectum. 2014 Mar;57(3):324-30. doi: 10.1097/DCR.0000000000000065. PMID 24509454
- [Background] Kingham TP, Pachter HL. Colonic anastomotic leak: risk factors, diagnosis, and treatment. J Am Coll Surg. 2009 Feb;208(2):269-78. doi: 10.1016/j.jamcollsurg.2008.10.015. Epub 2008 Dec 4. No abstract available. PMID 19228539
- [Background] Gorissen KJ, Benning D, Berghmans T, Snoeijs MG, Sosef MN, Hulsewe KW, Luyer MD. Risk of anastomotic leakage with non-steroidal anti-inflammatory drugs in colorectal surgery. Br J Surg. 2012 May;99(5):721-7. doi: 10.1002/bjs.8691. Epub 2012 Feb 9. PMID 22318712
- [Background] Ito M, Sugito M, Kobayashi A, Nishizawa Y, Tsunoda Y, Saito N. Relationship between multiple numbers of stapler firings during rectal division and anastomotic leakage after laparoscopic rectal resection. Int J Colorectal Dis. 2008 Jul;23(7):703-7. doi: 10.1007/s00384-008-0470-8. Epub 2008 Apr 1. PMID 18379795
- [Background] Kim JS, Cho SY, Min BS, Kim NK. Risk factors for anastomotic leakage after laparoscopic intracorporeal colorectal anastomosis with a double stapling technique. J Am Coll Surg. 2009 Dec;209(6):694-701. doi: 10.1016/j.jamcollsurg.2009.09.021. PMID 19959036
- [Background] Park JS, Choi GS, Kim SH, Kim HR, Kim NK, Lee KY, Kang SB, Kim JY, Lee KY, Kim BC, Bae BN, Son GM, Lee SI, Kang H. Multicenter analysis of risk factors for anastomotic leakage after laparoscopic rectal cancer excision: the Korean laparoscopic colorectal surgery study group. Ann Surg. 2013 Apr;257(4):665-71. doi: 10.1097/SLA.0b013e31827b8ed9. PMID 23333881
- [Background] Kawada K, Hasegawa S, Hida K, Hirai K, Okoshi K, Nomura A, Kawamura J, Nagayama S, Sakai Y. Risk factors for anastomotic leakage after laparoscopic low anterior resection with DST anastomosis. Surg Endosc. 2014 Oct;28(10):2988-95. doi: 10.1007/s00464-014-3564-0. Epub 2014 May 23. PMID 24853855
- [Background] Boni L, David G, Dionigi G, Rausei S, Cassinotti E, Fingerhut A. Indocyanine green-enhanced fluorescence to assess bowel perfusion during laparoscopic colorectal resection. Surg Endosc. 2016 Jul;30(7):2736-42. doi: 10.1007/s00464-015-4540-z. Epub 2015 Oct 20. PMID 26487209
- [Background] James DR, Ris F, Yeung TM, Kraus R, Buchs NC, Mortensen NJ, Hompes RJ. Fluorescence angiography in laparoscopic low rectal and anorectal anastomoses with pinpoint perfusion imaging--a critical appraisal with specific focus on leak risk reduction. Colorectal Dis. 2015 Oct;17 Suppl 3:16-21. doi: 10.1111/codi.13033. PMID 26394738
- [Background] Stergios K, Kontzoglou K, Pergialiotis V, Korou LM, Frountzas M, Lalude O, Nikiteas N, Perrea DN. The potential effect of biological sealants on colorectal anastomosis healing in experimental research involving severe diabetes. Ann R Coll Surg Engl. 2017 Mar;99(3):189-192. doi: 10.1308/rcsann.2016.0357. Epub 2016 Dec 5. PMID 27917665
- [Background] Lee S, Ahn B, Lee S. The Relationship Between the Number of Intersections of Staple Lines and Anastomotic Leakage After the Use of a Double Stapling Technique in Laparoscopic Colorectal Surgery. Surg Laparosc Endosc Percutan Tech. 2017 Aug;27(4):273-281. doi: 10.1097/SLE.0000000000000422. PMID 28614172
- [Background] Zhang L, Xie Z, Zhang W, Lin H, Lv X. Laparoscopic low anterior resection combined with "dog-ear" invagination anastomosis for mid- and distal rectal cancer. Tech Coloproctol. 2018 Jan;22(1):65-68. doi: 10.1007/s10151-017-1727-4. Epub 2017 Nov 28. No abstract available. PMID 29185063
- [Background] Chen ZF, Liu X, Jiang WZ, Guan GX. Laparoscopic double-stapled colorectal anastomosis without "dog-ears". Tech Coloproctol. 2016 Apr;20(4):243-7. doi: 10.1007/s10151-016-1437-3. Epub 2016 Feb 22. No abstract available. PMID 26902367
- [Background] D'Souza N, de Neree Tot Babberich MPM, d'Hoore A, Tiret E, Xynos E, Beets-Tan RGH, Nagtegaal ID, Blomqvist L, Holm T, Glimelius B, Lacy A, Cervantes A, Glynne-Jones R, West NP, Perez RO, Quadros C, Lee KY, Madiba TE, Wexner SD, Garcia-Aguilar J, Sahani D, Moran B, Tekkis P, Rutten HJ, Tanis PJ, Wiggers T, Brown G. Definition of the Rectum: An International, Expert-based Delphi Consensus. Ann Surg. 2019 Dec;270(6):955-959. doi: 10.1097/SLA.0000000000003251. PMID 30973385
- [Background] Factores asociados a la dehiscencia clínica de una anastomosis intestinal grapada: análisis multivariado de 610 pacientes consecutivos. Bannura et al. Rev. Chilena de Cirugía. Vol 58. Oct 2006; 341-346
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450